CLINICAL TRIAL: NCT06421701
Title: A Clinical Study of Anti-CD19 CAR-NK Cells in the Treatment of Refractory/Relapsed Systemic Lupus Erythematosus
Brief Title: Anti-CD19 CAR-NK Cells in Refractory/Relapsed Systemic Lupus Erythematosus
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-0530
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- anti-CD19 CAR-NK cells (Experimental): To evaluate the safety and efficacy of anti-CD19 CAR-NK cells in patients with refractory/relapsed systemic lupus erythematosus. All subjects will receive fludarabine/cyclophosphamide lymphodepletion followed by anti-CD19 CAR-NK cells infusion on Day 0, 3, and 6.
  Interventions: Drug: anti-CD19 CAR-NK cells

INTERVENTIONS:
Drug: anti-CD19 CAR-NK cells — Patients will receive Fludarabine and Cyclophosphamide for lymphodepletion conditioning. Anti-CD19 CAR-NK cells will be infused on Day 0, 3, and 6.

SUMMARY:
This study is a single-center, open-label, single-arm trial. The aim of this study is to investigate the safety and efficacy of anti-CD19 CAR-NK cells in patients with refractory/relapsed systemic lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up;
* Age range from 18 to 65 years old, regardless of gender;
* Fulfilling the 2019 ACR/EULAR classification criteria of SLE;
* Presence of anti-dsDNA or decreased C3/C4 levels;
* SLEDAI-2K≥8；
* Routine treatment is ineffective or the disease relapses after remission. Definition of routine treatment: use more than two drugs, including glucocorticoid (more than 1mg/kg/d), and any two or more of the following immunomodulatory drugs for more than 6 months: cyclophosphamide, mycophenolate mofetil, azathioprine, methotrexate, leflunomide, tacrolimus, ciclosporin, iguratimod, biological agents, including rituximab, belizumab, or telitacicept；
* Hemoglobin ≥ 80g/L; white blood cell count ≥ 3 × 10^9/L；neutrophil count ≥ 1.5 × 10^9/L; platelets ≥ 30 × 10^9/L;
* The functions of important organs are basically normal: ALT ≤ 2 × ULN; AST ≤ 2 × ULN; eGFR ≥ 30ml/min/1.73m2; total bilirubin ≤2.0 mg/dL; cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%; non-oxygenated blood oxygen saturation >94%; prothrombin time (PT) ≤ 1.5 × ULN；international standardized ratio (INR) ≤ 1.5 × ULN；
* Females of childbearing potential must use effective contraception during the study.

Exclusion Criteria:

* History of severe allergy or known hypersensitivity to any of the active ingredients of the cell product；
* Pregnant (or lactating) women;
* Severe lupus nephritis (defined as serum creatinine > 2.5 mg/dL or 221 μmol/L), treatment with hemodialysis within 8 weeks prior to screening；
* Other lupus crises, such as active central nervous system lupus, severe hemolytic anemia, severe thrombocytopenic purpura, severe agranulocytosis, severe myocardial damage, severe lupus pneumonia or pulmonary hemorrhage, severe lupus hepatitis, and severe vasculitis within 8 weeks prior to screening；
* Combined with other autoimmune diseases requiring systemic therapy except for secondary sjogren's syndrome;
* Clinically significant central nervous system diseases or pathological changes not caused by lupus prior to screening, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis;
* Abnormal test results for hepatitis B or C indicate the presence of an active or chronic infection, including positive HBsAg or positive HBcAb with HBV DNA levels exceeding the normal upper limit，positive hepatitis C antibody and detectable HCV RNA；positive serology for human immunodeficiency virus (HIV) or a known history of HIV infection; patients who test positive for HBsAg, have HBV DNA levels within the normal range, and are willing to reveive full-course antiviral therapy for hepatitis B are allowed to participate in this trial.
* Cytomegalovirus DNA levels in the peripheral blood exceeding the normal upper limits；
* Active or latent tuberculosis；
* Presence of uncontrollable bacterial, fungal, viral or other infections, requiring antibiotic therapy;
* Acquired and congenital immunodeficiency diseases；
* IgA deficiency;
* Other uncontrolled diseases: acute or chronic diseases that are clinically unstable or have not been effectively controlled and are not related to SLE；
* History of malignant diseases such as malignant tumors, except for adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, superficial bladder cancer, breast cancer;
* Any active skin disease that may interfere with the study assessment of SLE, including but not limited to psoriasis, dermatomyositis, systemic sclerosis, non-LE cutaneous lupus manifestations (eg, cutaneous vascular disease, periungual telangiectasia, fingertip sclerosis, rheumatoid nodules, erythema multiforme, leg ulcers) or drug-induced lupus；
* Prior treatment with cell therapy or any prior gene therapy product；
* Contraindication to cyclophosphamide in combination with fludarabine;
* Prior CD19-targeted therapy;
* Received live vaccine treatment within 4 weeks prior to screening;
* Subjects who have undergone major surgery within 8 weeks prior to screening, or who are scheduled to have surgery during the trial；
* Have received B-cell targeted therapy within 4 weeks prior to screening;
* Have received plasmapheresis within 3 months prior to screening;
* Have participated in other clinical studies within 3 months prior to screening;
* History of vital organ transplantation (eg, heart, lung, kidney, liver) or hematopoietic stem cell/or bone marrow transplantation；
* Situations in which investigators consider it inappropriate to participate in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects with adverse events | 12 months
  Incidence and severity of AEs and SAEs, including changes in laboratory values and vital signs as assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Proportion of subjects with Systemic Lupus Erythematosus Responder Index-4 (SRI-4) response | day 28, month 2, month 3, month 4, month 5, month 6, month 9 and month 12 after infusion.
  Proportion of patients with SRI-4 response: including SLEDAI-2000 ≥4-Point improvement, BILAG 2004 with no new A domain score AND no more than 1 new B domain scores, PGA with No worsening (<0.3-point increase).
Proportion of participants achieving definition of remission in SLE (DORIS) remission | day 28, month 2, month 3, month 4, month 5, month 6, month 9 and month 12 after infusion.
  The Definition of Remission in SLE (DORIS) is a standardized criterion to clearly define what constitutes remission in patients with systemic lupus erythematosus.
Proportion of participants achieving Lupus Low Disease Activity State (LLDAS) | day 28, month 2, month 3, month 4, month 5, month 6, month 9 and month 12 after infusion.
  The Lupus Low Disease Activity State (LLDAS) is a clinical treatment target designed for patients with systemic lupus erythematosus. It represents a state where the disease activity is kept at a low level, aiming to minimize symptoms and prevent long-term damage caused by the disease.
Changes in the Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2000) score from baseline | Within 12 months after anti-CD19 CAR-NK cell infusion
  Assessment of SLEDAI-2000 from baseline administration at various timepoints up to month 12 follow up visit.
Changes in the Physician Global Assessment (PGA) from baseline | Within 12 months after anti-CD19 CAR-NK cell infusion
  Assessment of PGA from baseline administration at various timepoints up to month 12 follow up visit.
Change in proteinuria measured by 24h proteinuria or urine protein creatinine ratio (UPCR) from baseline | Within 12 months after anti-CD19 CAR-NK cell infusion
  Assessment of 24h proteinuria or urine protein creatinine ratio (UPCR) from baseline administration at various timepoints up to month 12 follow up visit.
Changes in level of anti-nuclear antibody (ANA) in peripheral blood from baseline | Within 12 months after anti-CD19 CAR-NK cell infusion
  Assessment of ANA from baseline administration at various timepoints up to month 12 follow up visit.
Changes in levels of complement C3 and C4 in peripheral blood from baseline | Within 12 months after anti-CD19 CAR-NK cell infusion
  Assessment of C3 and C4 from baseline administration at various timepoints up to month 12 follow up visit.
CMAX of anti-CD19 CAR-NK cells | 12 months
  CMAX is defined as the highest concentration of anti-CD19 CAR-NK cell expansion in the peripheral blood.
TMAX of anti-CD19 CAR-NK cells | 12 months
  TMAX is defined as the time to reach the highest concentration of anti-CD19 CAR-NK cell expansion in the peripheral blood.

CONTACTS AND LOCATIONS:
Overall Officials: Huaxiang Wu, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University; Wenbin Qian, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, China, China

IPD SHARING:
Plan to Share IPD: No